CLINICAL TRIAL: NCT06183489
Title: A Multi-center, Open-label, Phase 2 Study of Elranatamab in Patients With High-risk Smoldering Multiple Myeloma
Brief Title: Use of Elranatamab in Patients With High-risk Smoldering Multiple Myeloma
Acronym: ERASMM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMN34/2023-505775-70-00
Record Dates: First submitted 2023-12-14; First posted 2023-12-27 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Smoldering Multiple Myeloma
Keywords: high-risk smoldering Multiple Myeloma; Elranatamab
MeSH Terms: conditions — Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Elranatamab (Experimental): Participant will receive elranatamab subcutaneously (SC) for 24 cycles (28-day cycle)
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — Elranatamab will be administered via a subcutaneous injection (SC)

SUMMARY:
This is a multicenter, single arm, open-label, Phase 2 study in high risk smoldering myeloma patients. The primary objective is to determine the efficacy of Elranatamab in patients with previously untreated high-risk SMM. The key-secondary objective is to determine the safety of Elranatamab in patients with previously untreated high-risk SMM.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Diagnosis of SMM for ≤5 years with measurable disease, defined as serum M protein:

   ≥1g/dL or urine M protein ≥200 mg/24 hours or involved serum FLC ≥100 mg/Land abnormal serum FLC ratio.
3. BMPCs ≥10% and <60%
4. Presence of at least 2 high risk factors, including

   1. Serum M protein ≥2 g/dL,
   2. BMPC >20%
   3. Serum involved/uninvolved FLC ratio > 20
5. ECOG performance status score of 0 or 1
6. Subjects must meet the following laboratory parameters, per laboratory reference range (performed at most 15 days before cycle 1 day 1)

   1. Absolute neutrophil count ≥1.0 x 109/L (ie, ≥1000/μL)
   2. Platelet count ≥75 x 109/L
   3. Aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN)
   4. Alanine aminotransferase (ALT) ≤2.5 x ULN
   5. Total bilirubin ≤1.5 x ULN, except in subjects with congenital bilirubinemia,such as Gilbert syndrome (in which case direct bilirubin ≤2.0 x ULN is required)
7. Subject must sign an informed consent form (ICF) or their legally acceptable representative must sign indicating that he or she understands the purpose of, and procedures required for the study and is willing to participate in the study.
8. Women of childbearing potential must have a negative serum or urine pregnancy test at screening and before starting study drug. They must commit to continued abstinence from heterosexual intercourse or begin 2 acceptable methods of birth control (One highly effective method and one additional effective method) used at the same time, and continuing for at least 5 months after the last dose of Elranatamab. Women must also agree to notify pregnancy during the study.

Exclusion Criteria:

1. Previous therapy with any systemic therapy for multiple myeloma.
2. Evidence of any of the following calcium, renal failure, anemia, bone lesions (CRAB) criteria or Myeloma Defining Events (SLiM CRAB) detailed below (attributable to the participants SMM involvement):

   1. Increased calcium levels: Corrected serum calcium >1 mg/dL above the ULN or >11 mg/dL
   2. Renal insufficiency: Determined by glomerular filtration rate (GFR) <40 mL/min/1.73 m² (Modification of Diet in Renal Disease [MDRD] Formula) or serum creatinine >2 mg/dL
   3. Anemia (hemoglobin 2 g/dL below lower limit of normal or <10 g/dL or both) transfusion support or concurrent treatment with erythropoietin stimulating agents is not permitted
   4. ≥ 1 bone lytic lesion
   5. BMPCs ≥60%
   6. Serum involved/uninvolved FLC ratio ≥100 and an involved FLC ≥100mg/L
   7. Whole body magnetic resonance imaging (WB-MRI) or positron emission tomography-computed tomography (PET-CT) with more than 1 bone focal lesion (≥5 mm in diameter)
3. Diagnosis of primary amyloidosis, POEMS syndrome, monoclonal gammopathy of undetermined significance, symptomatic multiple myeloma, or solitary plasmacytoma.
4. Subject has a diagnosis of Waldenström's macroglobulinemia, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
5. Subject has had plasmapheresis within 14 days of elegibility confirmation.
6. Myocardial infarction within 6 months prior to enrolment according to NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
7. Ongoing Grade 2 or higher peripheral sensory/motor peripheral neuropathy (PN), history of GBS or GBS variants, or history of grade 3 or higher peripheral motor polyneuropathy
8. Subject has had major surgery within 2 weeks before elegibility confirmation or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study.
9. Clinically relevant active infection or serious co-morbid medical conditions
10. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer free of disease since 5 years.
11. Female subject who is pregnant or breast-feeding
12. Serious medical or psychiatric illness likely to interfere with participation in study
13. Uncontrolled diabetes mellitus
14. Known HIV infection; Known active hepatitis B or C viral infection; known active COVID-19/SARS-CoV-2 infection
15. Live attenuated vaccine administered within 4 weeks of the first dose of study intervention
16. Ongoing treatment with corticosteroids : dose >10mg prednisone etc.
17. Person under guardianship, trusteeship or deprived of freedom by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Complete Remission (CR) rate | average 24 weeks
  Response of CR is defined as participants who achieve a CR or better (CR+sCR) according to IMWG response criteria, during the first 6 cycles of treatment and before a possible early termination of the treatment

SECONDARY OUTCOMES:
Overall response rate (ORR) | average 24 weeks
  Overall response rate (ORR) is defined as the proportion of participants achieving a confirmed PR or better according to the IMWG response criteria.
MRD-negative CR (MRD_CR) | average 24 weeks
  MRD-negative CR (MRD_CR) is defined as the proportion of participants achieving a MRD negativity (at or below the threshold of 10-5 by NGS) and CR or better according to the IMWG response criteria.
Progression-free survival (PFS) | time from the date of 1st dose to to the date of disease progression or death, assed up to 4 years after last dose
  defined as the time from the date of 1st dose of study drug to the date of first confirmed PD, as defined in the IMWG response criteria, or death due to any cause, whichever occurs first. If the participant is alive and w/o progression disease, the participant's data will be censored at the date of last disease assessment.
Time to progression (TTP) | time from the date of 1st dose to progression or death, assed up to 4 years after last dose
  Time to progression (TTP) is defined as the time from the date of 1st dose of study drug to the date of first documented PD, as defined in the IMWG response criteria. If the participant is w/o progression disease or die, the participant's data will be censored at the date of last disease assessment.
Progression free survival 2 (PFS2) | time from the date of 1st dose to progression on the next line of treatment or death,assed up to 4 years after last dose
  Progression free survival 2 (PFS2) is defined as the time from the date of 1st dose of study drug to the date of event, which is defined as death from any cause or PD as assessed by investigator that starts after the next line of therapy, whichever occurs first. If the participant starts next line of subsequent therapy without disease progression on study treatment, participant's data will be censored at the last disease assessment before starting next line of therapy. If participant starts next line of therapy after progression on study treatment and is still alive and not yet progress on next line of therapy, participant's data will be censored on the last date of follow-up.
Overall survival (OS) | time from the date of 1st dose to date of death, assed up to 4 years after last dose
  Overall survival (OS) is defined as the time from the date of 1st dose of study drug to the date of death. If the participant is alive, the participant's data will be censored at the date the participant was last known to be alive
Time to response (TTR) | time frrom the date of 1st dose to the first documented response
  Time to response (TTR) is defined as the time from the date of 1st dose of study drug to the first documented response (≥PR). If the participant is alive, w/o progression disease and w/o documented response (≥PR), the participant's data will be censored at the date of last disease assessment. If the participant have a progression or die before a documented response (≥PR), the participant's data will have a competing event at the date of PFS event.
Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core module (EORTC QLQ-C30) | from screening, cycle 1 and every 3 cycles there after up to end of treatment and 28 days after last treatment
  The EORTC QLQ-C30 is a 30-item questionnaire containing both single and multi-item measures. These include five functional scales (Physical, Role, Cognitive, Emotional, and Social Functioning), three symptom scales (Fatigue, Pain, and Nausea/Vomiting), a Global Health Status/ Quality-of-Life (QoL) scale, and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). The scores ranges from 0-100, a high score for functional scales and for Global Health Status/QoL represent better functioning ability or Health-Related Quality-ofLife (HRQoL), whereas a high score for symptom scales and single items represents significant symptomatology.
Change in EORTC QLQ- 20-item Multiple Myeloma module (MY-20) score | from screening, cycle 1 and every 3 cycles there after up to end of treatment and 28 days after last treatment
  The EORTC QLQ-MY20 is a supplement to the QLQ-C30 instrument used in subjects with MY. The module comprises 20 questions that address four myeloma-specific HRQoL domains: Disease Symptoms, Side Effects of Treatment,Future Perspective, and Body Image. A high score for Disease Symptoms and Side Effects of Treatment represents a high level of symptomatology or problems, whereas a high score for Future Perspective and Body Image represents better outcomes.

CONTACTS AND LOCATIONS:
Locations (25):
- Helsinki University Hospital, Helsinki, Finland
- France (7):
  - CHD Vendée, La Roche-sur-Yon
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - CHU Saint Eloi Département d'Hématologie Clinique, Montpellier
  - CHU Hôtel-Dieu, 1, place Alexis Ricordeau, 44093 NANTES Cedex 1, FRANCE, Nantes
  - CHU NICE - Hôpital Archet, Nice
  - CHU Poitiers - Pôle régional de Cancérologie, Poitiers
  - CHRU Hôpital Bretonneau, Tours
- Alexandra General Hospital -Department of Clinical Therapeutics N.K. Univ. of Athens, Athens, Greece
- Italy (12):
  - AOU Consorziale Policlinico di Bari, Bari
  - A.O. Papa Giovanni XXIII, Bergamo
  - A.O.U. Careggi, Florence
  - A.O.U. Policlinico S. Martino - Ematologia, Genova
  - Meldola-Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola
  - Ospedale Papardo, Messina
  - A.O.U. Maggiore della Carità Novara, Novara
  - A.O. di Padova, Padua
  - A.O.U. di Parma - U.O Ematologia e CTMO, Parma
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Ospedale Santo Spirito Ospedale -Azienda Sanitaria Locale Di Pescara, Roma
  - Clinica Ematologica Azienda Sanitaria Universitaria Friuli Centrale, Udine
- Netherlands (3):
  - Maastricht UMC, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC, Rotterdam
- Oslo Myeloma Center, Oslo, Norway